CLINICAL TRIAL: NCT02501603
Title: An Open-label, Multicenter Phase II Study of Afatinib Plus Weekly Taxol as Second Line Treatment for Advanced/Recurrent Gastric and Gastroesophageal Junction Cancer
Brief Title: Afatinib, Paclitaxel, 2nd Line, Advanced Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Sun Young Rha, Professor, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2015-0244
Record Dates: First submitted 2015-07-08; First posted 2015-07-17 (Estimated); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Afatinib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- afatinib plus paclitaxel (Experimental): afatinib plus paclitaxel
  Interventions: Drug: afatinib; Drug: paclitaxel

INTERVENTIONS:
Drug: afatinib — Afatinib 40mg daily oral administration
Drug: paclitaxel — Paclitaxel 80mg/m2 IV weekly (day 1,8,15)

SUMMARY:
For the gastric cancer, paclitaxel is recommended as salvage standard treatment. Afatinib is a novel, potent, small ErbB family blocker that covalently binds and irreversibly blocks signaling through activated EGFR, HER2 and ErbB4 receptors, as well as the transphosphorylation of ErbB3. The investigators suggest a randomized phase II trial of afatinib plus weekly taxol(paclitaxel) for previously treated EGFR positive gastric cancer patients. The aim of current trial is to evaluate the antitumor efficacy of afatinib for target enriched patients in gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed locally advanced or metastatic gastric cancer and gastroesophageal junction cancer
2. EGFR 2+ or 3+ expression (immunohistochemistry)
3. ECOG performance status of 0 to 1
4. Male or female; ≥ 19 years of age
5. Documented disease progression after one prior therapy, in locally advanced or metastatic setting
6. patients received last adjuvant chemotherapy less than six months can be enrolled into this study
7. Her2 positive patients must be progressed after prior trastuzumab based chemotherapy
8. Subjects with measurable lesion (using RECIST 1.1 criteria)
9. Subjects who meet the following criteria:

   * Absolute neutrophil count (ANC) ≥ 1000 /µL (*ANC = Neutrophil segs ＋ Neutrophil bands)
   * Platelet count ≥ 80,000/ µL
   * Serum creatinine < 1.5 x upper limit of normal (ULN) or Creatinine clearance ≥50 mL/min using Cockcroft, Gault method
   * AST (SGOT) and ALT (SGPT) : 3 x upper limit of normal (ULN) (If there is Liver Metastasis : 5 x upper limit of normal (ULN))
   * Total bilirubin : 1.5 x upper limit of normal (ULN)
10. Provision of written informed consent prior to any study procedure

Exclusion Criteria:

1. Any unresolved chronic toxicity greater than CTC grade 2 from previous anticancer therapy.
2. Any previous chemotherapy or immunotherapy within 2 weeks
3. Any major operation or irradiation within 4 weeks of baseline disease assessment
4. Two or more previous systemic cytotoxic chemotherapy (adjuvant chemotherapy is not counted)
5. Any clinically significant gastrointestinal abnormalities which may impair intake or absorption of the study drug
6. Previously taxol(paclitaxel)-exposed patients
7. Subjects with symptomatic central nervous system (CNS) metastases who are neurologically unstable or have required increasing doses of steroids within the 2 weeks prior to study entry to manage CNS symptoms
8. Other co-existing malignancies or malignancies diagnosed within the last 3 years with the exception of basal cell carcinoma, thyroid cancer or cervical cancer in situ.
9. Subjects with an uncontrolled major cardiovascular disease (including AMI within 12 months, unstable angina within 6 months, over NYHA class III congestive heart failure, congenital long QT syndrome, 2° or more AV Block and uncontrolled hypertension)
10. Pregnant or lactating female
11. Patients with contraindicated medication
12. History of interstitial lung disease (ILD) or presence of ILD on chest X-ray
13. Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2016-07; Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
compare progression free survival as measured by RECIST 1.1 | Every 6 weeks until progression, an expected average of 10 months
  To identify antitumor activity of afatinib plus weekly taxol(paclitaxel) and explore predictive biomarker

SECONDARY OUTCOMES:
antitumor efficacy as measured by RECIST 1.1 | every 6 weeks until progression, an expected average of 10 months
safety as measured by CTCAE | every 3 weeks until progression, an expected average of 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Sun Young Rha, Principal Investigator — Severance Hospital, Yonsei University Health System, Yonsei Cancer Center
Locations (1):
- Severance Hospital, Yonsei University Health System, Yonsei Cancer Center, Seoul, South Korea